CLINICAL TRIAL: NCT03269292
Title: Clinical Characteristics and Treatment Outcomes of Patients With Autoimmune Hemolytic Anemia in Assiut University Hospital
Brief Title: Clinical Characteristics and Treatment Outcomes of Patients With Autoimmune Hemolytic Anemia
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehab A. Abdelmenam, Principal Investigator, Assiut University
Other Study IDs: AIHA in assiut
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- warm autoimmune hemolytic anemia: corticosteroid either oral form or intravenous followed by oral

SUMMARY:
Autoimmune hemolytic anemia is characterized by shortened red blood cell survival and a positive Coombs test. The responsible autoantibodies may be either warm reactive or cold reactive. The rate of hemolysis and the severity of the anemia may vary from mild to severe and life-threatening. Diagnosis is made in the laboratory by the findings of anemia, reticulocytosis, a positive Coombs test, and specific serologic tests. The prognosis is generally good but renal failure and death sometimes occur, especially in cases mediated by drugs.

DETAILED DESCRIPTION:
Hemolysis is the premature destruction of erythrocytes. A hemolytic anemia will develop if bone marrow activity cannot compensate for the erythrocyte loss. The severity of the anemia depends on whether the onset of hemolysis is gradual or abrupt and on the extent of erythrocyte destruction Hemolysis can be due to hereditary and acquired disorders. Acquired causes of hemolysis include immune disorders, Toxic chemicals and drugs, Antiviral agents and Physical damage .

Autoimmune hemolytic anemia (AIHA) exhibits two important characteristics: shortened red blood cell (RBC) survival and presence of autoantibodies directed toward autologous RBCs, usually demonstrated by a positive direct antiglobulin (Coombs) test (DAT). AIHA is classified by the temperature at which autoantibodies bind optimally to RBCs. In warm antibody AIHA, which constitutes about 80-90% of adult cases, hemolysis is mediated by antibodies which bind to RBCs at 37 °C (98.6 °F. In cryopathic hemolytic syndromes, cold-reactive autoantibodies exhibit affinity for RBCs optimally at temperatures below body temperature. In adults, most of the cold-reactive antibodies are agglutinins of the immunoglobulin M (IgM) isotype. In children, cold hemolysins (generally IgG) are most common. Unusual patients with mixed AIHA exhibit both cold-reactive and warm-reactive autoantibodies .

Each of these types of AIHA may be sub-classified based on the presence or absence of underlying diseases. In the absence of an underlying disease, the AIHA is termed primary or idiopathic. When AIHA occurs as a manifestation or complication of another disease, the term secondary AIHA is used. Chronic lymphocytic leukemia (CLL) and lymphomas account for about half of all secondary AIHA cases. Systemic lupus erythematosus (SLE) and other autoimmune diseases also account for a large number of secondary AIHA cases. Certain drugs also mediate immune injury to RBCs. Three mechanisms are recognized and two of these involve elements of autoimmunity, in which autoantibodies recognize and bind to specific RBC epitopes in concert with drugs or their metabolites or in which the autoantibody binds to RBC epitopes without the presence of drug

Diagnosis The signs and symptoms of AIHA are nonspecific and common to all types of anemia . The primary symptoms include exertional dyspnea, dyspnea at rest, varying degrees of fatigue, and signs and symptoms of the hyperdynamic state, such as bounding pulses, palpitations…etc

The laboratory findings of drug-induced AIHA may resemble those of warm antibody AIHA or a cryopathic hemolytic syndrome, depending on the mechanism of the autoantibody induction and the target antigen. A high index of suspicion on the part of the clinician and discussions with blood bank personnel can usually reveal the role of the drug.

complete blood count Peripheral blood smear : This test can detect an anemia, pancytopenia, and infections. Along with the differential count, a complete blood count can help diagnose hematologic malignancies and other hematological disorders. The platelet count usually is normal in most hemolytic anemias.

An increased reticulocyte count represents increased RBC production and is a criterion for hemolysis but is not specific for hemolysis. Thrombocytopenia associated with positive direct coombs test occur in evans syndrome .

Serum lactate dehydrogenase (LDH) study : Serum LDH elevation is a criterion for hemolysis, but is not specific

Serum haptoglobin : A low serum haptoglobin level is a criterion for moderate-to-severe hemolysis.

Indirect bilirubin : Unconjugated bilirubin is a criterion for hemolysis, but it is not specific , the level of indirect bilirubin usually is less than 3 mg/dL.

Direct antiglobulin test (DAT):

The DAT result is usually positive in autoimmune hemolytic anemia (AIHA), but it may occasionally be negative in this disorder. DAT-negative AIHAs have been reviewed. From 5-10% of all AIHAs are DAT negative. The polybrene test can detect DAT-negative AIHA.

Treatment all of the drugs used in the treatment of AIHA are largely or partly directed against the patient's natural immune system, which may, in turn, extensively derail the immune system due to treatment. .The first-line therapy for warm AIHA are corticosteroids, which are effective in 70-85% of patients and should be slowly tapered over a time period of 6-12 months. For refractory/relapsed cases, the current sequence of second-line therapy is splenectomy (effective approx. in 2 out of 3 cases but with a presumed cure rate of up to 20%), rituximab (effective in approx. 80-90% of cases), and thereafter any of the immunosuppressive drugs (azathioprine, cyclophosphamide, cyclosporin, mycophenolate mofetil). Additional therapies are intravenous immunoglobulins, danazol, plasma-exchange, and alemtuzumab and high-dose cyclophosphamide as last resort option. As the experience with rituximab evolves, it is likely that this drug will be located at an earlier point in therapy of warm AIHA, before more toxic immunosuppressants, and in place of splenectomy in some cases. In coronary artery disease , rituximab is now recommended as first-line treatment

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed warm auto Immune hemolytic anemia primary or secondary(CLL, Lymphoma, rheumatoid arthritis

, SLE,Drug-induced )

Exclusion Criteria:

1. All types of congenital hemolytic anemia
2. Microangiopathic hemolytic anemia ( Thrombotic thrombocytopenic purpura (TTP) , Hemolytic-uremic syndrome (HUS) , Disseminated intravascular coagulation (DIC) )
3. Alloimmune hemolytic anemia
4. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients above 18 years or more diagnosed AIHA at Assiut university hospital
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin | three week from baseline
  Efficacy endpoint assesment
frequency of drug-related side effects | three week from base line
  safety endpoint

SECONDARY OUTCOMES:
Dose of steroid treatment | at 3 weeks, three months, six month, one year from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Essam Abdel Monem El-beih, professor, Study Director — Assiut University; wael ahmed abbas, professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Result] Packman CH. The Clinical Pictures of Autoimmune Hemolytic Anemia. Transfus Med Hemother. 2015 Sep;42(5):317-24. doi: 10.1159/000440656. Epub 2015 Sep 11. PMID 26696800
- [Result] Dhingra KK, Jain D, Mandal S, Khurana N, Singh T, Gupta N. Evans syndrome: a study of six cases with review of literature. Hematology. 2008 Dec;13(6):356-60. doi: 10.1179/102453308X343518. PMID 19055865
- [Result] Garratty G. Immune hemolytic anemia associated with negative routine serology. Semin Hematol. 2005 Jul;42(3):156-64. doi: 10.1053/j.seminhematol.2005.04.005. PMID 16041665
- [Result] Kamesaki T, Oyamada T, Omine M, Ozawa K, Kajii E. Cut-off value of red-blood-cell-bound IgG for the diagnosis of Coombs-negative autoimmune hemolytic anemia. Am J Hematol. 2009 Feb;84(2):98-101. doi: 10.1002/ajh.21336. PMID 19105232
- [Result] Zanella A, Barcellini W. Treatment of autoimmune hemolytic anemias. Haematologica. 2014 Oct;99(10):1547-54. doi: 10.3324/haematol.2014.114561. PMID 25271314
- [Result] Michel M. [Characteristics of warm autoimmune hemolytic anemia and Evans syndrome in adults]. Presse Med. 2008 Sep;37(9):1309-18. doi: 10.1016/j.lpm.2008.01.026. Epub 2008 Jul 17. French. PMID 18644324
- [Result] Salama A. Treatment Options for Primary Autoimmune Hemolytic Anemia: A Short Comprehensive Review. Transfus Med Hemother. 2015 Sep;42(5):294-301. doi: 10.1159/000438731. Epub 2015 Aug 10. PMID 26696797